CLINICAL TRIAL: NCT03286114
Title: Augmentation of the Graft vs. Leukemia Effect Via Checkpoint Blockade With Pembrolizumab for Relapse of Primary Malignancy After Allogeneic Hematopoietic Stem Cell Transplant: A Feasibility Study
Brief Title: Augmentation of the Graft vs. Leukemia Effect Via Checkpoint Blockade With Pembrolizumab
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of patient population
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2017.056; HUM00129255 (Other: University of Michigan)
Record Dates: First submitted 2017-09-08; First posted 2017-09-18 (Actual); Results first posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-04

CONDITIONS: Myelodysplastic Syndromes; Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Pembrolizumab (Experimental)
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — 200mg IV every 21 days
  Other Names: KEYTRUDA

SUMMARY:
This is a single arm, open-label, Phase 1b study of pembrolizumab for patients with myelodysplastic syndrome (MDS), acute myeloid leukemia (AML), and acute lymphoblastic leukemia (ALL) whose disease has relapsed after receiving allogeneic hematopoetic stem cell transplant.

ELIGIBILITY:
Inclusion Criteria:

* Acute Myeloid Leukemia (AML), Acute Lymphoblastic Leukemia (ALL) or Myelodysplastic Syndrome (MDS) in confirmed relapse
* Confirmation of 'measurable disease'
* Patient may not have received definitive salvage chemotherapy for their post-transplant relapse within the past 21 days.
* Be willing and able to provide written informed consent/assent for the trial
* Be ≥ 18 years of age on day of signing informed consent
* Be willing to provide tissue from bone marrow biopsies
* Have a performance status of 0, to 1 on the ECOG Performance Scale. Eastern Cooperative Oncology Group Performance Status: an attempt to quantify cancer patients' general well-being and activities of daily life. The score ranges from 0 to 5 where 0 is asymptomatic and 5 is death.
* Demonstrate adequate organ function
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication.
* Female subjects of childbearing potential must be willing to use an adequate method of contraception
* Male subjects of childbearing potential must agree to use an adequate method of contraception

Exclusion Criteria:

* Has had relapse prior to primary neutrophil engraftment or ≤21 days post HCT.
* Has received >1 line of chemotherapy or other treatment directed towards post-transplant relapse prior to study entry
* Rapidly progressive relapse requiring urgent chemotherapy as determined by treating physician
* Is currently participating and receiving study therapy of an investigational agent and received study therapy within 2 weeks of the first dose of treatment.
* Has a diagnosis of active GvHD (≥ Grade I)
* Receiving systemic steroid therapy of > 10mg prednisone daily or equivalent*
* Has received GM-CSF within 14 days of first dose of pembrolizumab
* Has a known history of active TB (Bacillus Tuberculosis)Hypersensitivity to pembrolizumab or any of its excipients
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered from adverse events
* Has had prior chemotherapy within 21 days or radiation therapy within 14 days prior to study Day 1 or who has not recovered from adverse events
* Has a known additional (secondary) malignancy that is progressing or requires active treatment
* Has known or suspected active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has a history of (non-infectious) pneumonitis that required steroids, or current pneumonitis
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent
* Has a known history of Human Immunodeficiency Virus (HIV)
* Has known active Hepatitis B or Hepatitis C
* Has received a live vaccine within 30 days of planned start of study therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2020-10-22 (Actual); Study Completion 2021-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Magenau, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Magenau JM, Frame DG, Riwes M, Maciejewski J, Anand S, Pawarode A, Perry AM, Geer M, Braun T, Ghosh M, Reddy P. PD-1 inhibition for relapse after allogeneic transplantation in acute myeloid leukemia and myelodysplastic syndrome. Blood Adv. 2025 Aug 12;9(15):3878-3886. doi: 10.1182/bloodadvances.2024015200. PMID 40198769

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pembrolizumab
Started | 16
Completed | 7
Not Completed | 9
Not completed — Adverse Event | 6
Not completed — Death | 3

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients That Demonstrate Clinical Benefit From Treatment
Description: This study will assess if the study drug is promising for further study. The study drug will be considered promising if at least 4 patients receive a clinical benefit or if any complete response is seen. Clinical benefit is defined as either stable disease, partial remission or complete remission to treatment.
  Complete remission (CR) will be defined as achieving a morphologic leukemia free state by achieving all of the following criteria: bone marrow myeloblasts < 5% by morphologic assessment; AND absence of circulating blasts with phenotypic or morphologic features of leukemia (e.g. Auer rods) AND no evidence of extramedulary disease.
  Partial remission (PR) will be defined as a ≥ 50% reduction in bone marrow blast percentage to 5-25% or marrow blasts < 5% with persistent Auer rods, flow cytometric or cytogenetic disease.
  SD will be defined as ≤ 5% increase in blasts or decreased blast percentage in the bone marrow that does not meet the criteria for PR.
Time Frame: Day 77
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 16
Participants | 6

2. Primary Outcome: The Number of Patients That Respond to Treatment
Description: This study will assess the number of patients that respond to treatment by overall response rate (ORR). ORR is defined as the number of patients will complete remission and partial remission.
  Complete remission (CR) will be defined as achieving a morphologic leukemia free state by achieving all of the following criteria: bone marrow myeloblasts < 5% by morphologic assessment; AND absence of circulating blasts with phenotypic or morphologic features of leukemia (e.g. Auer rods) AND no evidence of extramedulary disease.
  Partial remission (PR) will be defined as a ≥ 50% reduction in bone marrow blast percentage to 5-25% or marrow blasts < 5% with persistent Auer rods, flow cytometric or cytogenetic disease.
Time Frame: Day 77
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 16
Participants | 3

3. Primary Outcome: Graft Versus Host Disease (GvHD) or Other Significant Immune Mediated Toxicities
Description: The number of patients that experience Graft Versus Host Disease (GvHD) or other significant immune mediated toxicities
Time Frame: 30 Days Post Treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 16
Participants
  GVHD | 9
  mmune-related SAEs | 2

4. Secondary Outcome: Overall Survival
Description: The number of patients alive at 1 year
Time Frame: 1 Year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 16
percentage of participants | 37.5 [15.4 to 59.8]

5. Secondary Outcome: Event- Free Survival
Description: The number of patients alive at 1 year without disease
Time Frame: 1 Year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 16
percentage of participants | 31.3 [11.1 to 53.7]

ADVERSE EVENTS:
Time Frame: All adverse event data (serious and non-serious) collected from the time of the initial study treatment administration through 30 days after the last dose of study treatment. An average of 3 months.
Arm/Group | Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 12/16
Serious Adverse Events (participants affected / at risk) | 16/16
Other Adverse Events (participants affected / at risk) | 6/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=16)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (2)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 7 (7)
Fever (General disorders) | 2 (2)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Hyponatremia (Investigations) | 1 (1)
Lung infection (Infections and infestations) | 2 (2)
Mucositis oral (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3)
Sepsis (Infections and infestations) | 2 (2)
Syncope (Cardiac disorders) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Immune system disorders - Other, specify (Immune system disorders) | 5 (5) — GVHD - Gut
Immune system disorders - Other, specify (Immune system disorders) | 3 (3) — GVHD - Liver
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) — Bacteremia
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) — Infectious Colitis
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) — Fungal Infection
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=16)
Alanine aminotransferase increased (Investigations) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Blood bilirubin increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Investigations) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Immune system disorders - Other, specify (Immune system disorders) | 2 (2) — GVHD - Skin

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-16): https://cdn.clinicaltrials.gov/large-docs/14/NCT03286114/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-19): https://cdn.clinicaltrials.gov/large-docs/14/NCT03286114/ICF_001.pdf